CLINICAL TRIAL: NCT03581760
Title: Effect of a Cycling Exercise on Restoration of Muscle Strength in Patients Undergoing Mechanical Ventilation
Brief Title: Cycling Exercise in Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KARIM-08-Motomed; MH CZ - DRO-FNOs/2017 (Other Grant/Funding Number: Ministry of Health of the Czech Republic)
Record Dates: First submitted 2018-06-12; First posted 2018-07-10 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Muscle Weakness; Mechanical Ventilation Complication
Keywords: cycling exercise; mechanically ventilated patient; muscle strength assessment; muscle weakness
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Intervention Model Description: Patients enrolled in the study will be randomized into two groups - active intervention and control group.
Masking Description: This is an open-label study, no masking model is applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cycling Exercise (Experimental): Patients randomized into this arm will undergo cycling exercise once a day while on mechanical ventilation at intensive care unit.
  Interventions: Other: Cycling Exercise; Other: Conventional Physiotherapy
- Conventional Physiotherapy (Active Comparator): Patients randomized into this arm will undergo conventional physiotherapy twice a day while on mechanical ventilation at intensive care unit.
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Other: Cycling Exercise — Cycling exercise will be performed in the patients once a day.
  Arms: Cycling Exercise
Other: Conventional Physiotherapy — Conventional physiotherapy will be performed in the patients twice a day.

SUMMARY:
Prolonged critical illness renders survivors with increased long-term morbidity associated with high healthcare costs. Muscle weakness and fatigue are reported as the main contributors to long-term poor functional outcomes. Emerging evidence for early mobilisation demonstrates reduction in the number of ventilator days and hospital length of stay. It has been demonstrated that daytime motoring (passive and active) can improve functional capacity in intensive care patients. The aim of the proposed study is to evaluate the effect of cycling exercise in patients on mechanical ventilation appointed to weaning process.

DETAILED DESCRIPTION:
This prospective randomized study is being performed at the Department of Anesthesiology, Resuscitation and Intensive Care (CARIM) of the University Hospital Ostrava.

All mechanically ventilated patients are followed. At the time of weaning initiation, the randomization into two groups (the study (cycling) and control group) is performed. The physiotherapy will be carried out twice a day in both groups according to the mobility protocol. The cycling exercise is performed only in the study group, once a day. Before a patient is released from the ICU, a cycling test, dynamometry test will be performed on both groups.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* ICU admission
* Mechanically ventilated for more than 5 days
* Indications for starting weaning
* Informed consent for participation

Exclusion Criteria:

* Inability to use cycling exercise: trauma or operation of lower limbs, pelvis, open abdomen, non-cooperation (qualitative and quantitative disturbance of consciousness)
* Encephalopathy (ischemic, traumatic)
* Extreme obesity (body mass index ≥ 40)
* Anticipated survival time ≤ 7 days
* Patient height ≤ 1.5 m
* More than 48 hours of mechanical ventilation outside of the department

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Number of ventilator days | 43 months
  The influence of cycling exercises on the number of ventilator days will be assessed in the patients. The number of ventilator days will be compared in both groups of patients.

SECONDARY OUTCOMES:
Muscle strength | 43 months
  Muscle strength will be assessed in the mechanically ventilated patients in both groups on the Medical Research Council Manual Muscle Testing scale. This muscle scale grades muscle power on a scale of 0 to 5 in relation to the maximum expected for that muscle; the higher the measured value, the bigger the muscle strength and vice versa.

CONTACTS AND LOCATIONS:
Overall Officials: Renáta Zoubková, PhDr., Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
The investigators have not decided to share the IPD with other researchers.

REFERENCES:
- [Background] Bailey P, Thomsen GE, Spuhler VJ, Blair R, Jewkes J, Bezdjian L, Veale K, Rodriquez L, Hopkins RO. Early activity is feasible and safe in respiratory failure patients. Crit Care Med. 2007 Jan;35(1):139-45. doi: 10.1097/01.CCM.0000251130.69568.87. PMID 17133183
- [Background] Morris PE, Goad A, Thompson C, Taylor K, Harry B, Passmore L, Ross A, Anderson L, Baker S, Sanchez M, Penley L, Howard A, Dixon L, Leach S, Small R, Hite RD, Haponik E. Early intensive care unit mobility therapy in the treatment of acute respiratory failure. Crit Care Med. 2008 Aug;36(8):2238-43. doi: 10.1097/CCM.0b013e318180b90e. PMID 18596631
- [Background] Schweickert WD, Pohlman MC, Pohlman AS, Nigos C, Pawlik AJ, Esbrook CL, Spears L, Miller M, Franczyk M, Deprizio D, Schmidt GA, Bowman A, Barr R, McCallister KE, Hall JB, Kress JP. Early physical and occupational therapy in mechanically ventilated, critically ill patients: a randomised controlled trial. Lancet. 2009 May 30;373(9678):1874-82. doi: 10.1016/S0140-6736(09)60658-9. Epub 2009 May 14. PMID 19446324
- [Background] Morris PE, Griffin L, Berry M, Thompson C, Hite RD, Winkelman C, Hopkins RO, Ross A, Dixon L, Leach S, Haponik E. Receiving early mobility during an intensive care unit admission is a predictor of improved outcomes in acute respiratory failure. Am J Med Sci. 2011 May;341(5):373-7. doi: 10.1097/MAJ.0b013e31820ab4f6. PMID 21358312
- [Background] Burtin C, Clerckx B, Robbeets C, Ferdinande P, Langer D, Troosters T, Hermans G, Decramer M, Gosselink R. Early exercise in critically ill patients enhances short-term functional recovery. Crit Care Med. 2009 Sep;37(9):2499-505. doi: 10.1097/CCM.0b013e3181a38937. PMID 19623052